CLINICAL TRIAL: NCT04430647
Title: Phaco-UCP; Combined Phacoemulsification and Ultrasound Ciliary Plasty Versus Phacoemulsification Alone for Management of Coexisting Cataract and Open Angle Glaucoma
Brief Title: Phaco-UCP Versus Phaco Alone for OAG and Cataract
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ameera Gamal Abdelhameed (Other)
Collaborators: Dar Alshifa hospital Kuwait (Unknown)
Responsible Party: Sponsor-Investigator, Ameera Gamal Abdelhameed, Lecturer of Ophthalmology, Mansoura University
Organization: Mansoura University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Phaco-UCP in OAG and cataract
Record Dates: First submitted 2020-06-09; First posted 2020-06-12 (Actual); Last update posted 2020-06-12 (Actual); Status verified 2020-06

CONDITIONS: Cataract; Glaucoma, Open-Angle
MeSH Terms: conditions — Cataract; Glaucoma, Open-Angle | interventions — Phacoemulsification

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- phaco-UCP (Experimental): Under peribulbar anesthesia, UCP was performed first, followed by phacoemulsification. UCP was performed using the same technique described before [18]. For all treatments, 2nd generation probe was used (EyeOP1, Eye Tech care; France) with the same parameters; Operating frequency was 21 MHz. Number of sectors activated was 6. Acoustic power was 2.45 W; duration of each shot was 8s; and the time between shots was 20s. The probe diameter (11, 12 or 13 mm) was determined according to the eye's biometric readings. The coupling cone was centered on the eye and kept in place with low vacuum suction, followed by introduction of the treatment probe inside the cone, then activation of the transducers by constantly pressing the foot switch. Once UCP treatment was finished, phacoemulsification was commenced
  Interventions: Procedure: combined phacoemulsification and ultrasound ciliary plasty (Phaco-UCP)
- Phaco alone (Active Comparator): A standard phacoemulsification was performed with 2.2 mm clear corneal incision, continuous curvilinear capsulorhexis, phacoemulsification and intrabagal implantation of foldable acrylic intraocular lens (AcrySof® IQ SN60WF monofocal; Alcon Laboratories Inc, Fort Worth, TX, USA) for all patients. Irrigation-aspiration was performed for at least 30 seconds to remove any viscoelastic from the anterior chamber. Reformation of the anterior chamber was done with balanced saline solution (BSS), followed by hydration of the corneal wound and side port.
  Interventions: Procedure: Phacoemulsification alone

INTERVENTIONS:
Procedure: combined phacoemulsification and ultrasound ciliary plasty (Phaco-UCP) — performing ultrasound ciliary plasty then performing standard phacoemulsification
  Arms: phaco-UCP
Procedure: Phacoemulsification alone — standard phacoemulsification for catarct extraction
  Arms: Phaco alone

SUMMARY:
This study was carried out to evaluate the safety and efficacy of combined phacoemulsification and Ultrasound ciliary plasty (Phaco-UCP) as a first-line surgical treatment of coexisting cataract and op

/en angle glaucoma compared to phacoemulsification alone. To our knowledge, this is the first report of results of combined Phaco-UCP

DETAILED DESCRIPTION:
the study involved 61 eyes of 61 patients with coexisting cataract and open angle glaucoma, 31 eyes were managed with Phaco-UCP and 30 eyes of age and sex matched patients were managed with phacoemulsification alone.

Patients were randomized for either combined phacoemulsification and ultrasound ciliary plasty (Phaco-UCP) (the study group) or phacoemulsification alone (the control group). All surgeries were performed by one experienced surgeon (Y EZ).

Preoperative evaluation included manifest refraction, BCVA measurement, slit-lamp biomicroscopy, gonioscopy, indirect ophthalmoscopy, measurement of IOP with Goldmann applanation tonometry (average of 3 readings taken). Corneal diameter (White-to-white) and axial length measurement were done using IOL Master 500 (Carl Zeiss Meditec AG., Germany). Ultrasound pachymetry with Tomey SP-100 (Tomey Corp. Nagoya, Japan) and visual fields using Humphrey Field Analyzer (24-2, SITA, standard program Carl Zeiss Meditec AG., Germany) were also performed.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with POAG or pseudoexfoliation glaucoma with coexisting visually significant cataract that required phacoemulsification

Exclusion Criteria:

* patients with any other type of glaucoma, including narrow angle glaucoma, neovascular, uveitic or angle recession glaucoma, patients with advanced glaucoma characterized by advanced optic disc cupping or visual field damage, history of glaucoma or intraocular surgery and other ocular diseases that would affect safety or interfere with the procedure. We also excluded patients with incomplete follow-up or missing data

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
reduction in intraocular pressure | 18 months postoperative
  Qualified Success was defined as an IOP reduction of at least 20 % from baseline value, with an IOP that is between 6 - 21 mm Hg, without the need for additional antiglaucoma medications or glaucoma surgery
reduction in r the number of antiglaucoma medications. | 18 months postoperative
  reduction of the number of antiglaucoma medication or at least no increase in the number

SECONDARY OUTCOMES:
BCVA improvement | 18 months postoperative
  improvement of best corrected visual acuity
intraoperative and postoperative complications. | intraoperative and 18 months postoperative
  hyphema or vitreous hemorrhage necessitating surgical intervention, choroidal hemorrhage, chronic uveitis, endophthalmitis, hypotony (IOP ≤ 5 mm Hg), phthisis, IOL dislocation, and retinal detachment.

CONTACTS AND LOCATIONS:
Overall Officials: Magda Torky, MD, Principal Investigator — Mansoura University
Locations (1):
- Mansoura University, Al Mansurah, Dakahlia Governorate, Egypt

REFERENCES:
- [Background] Pascolini D, Mariotti SP. Global estimates of visual impairment: 2010. Br J Ophthalmol. 2012 May;96(5):614-8. doi: 10.1136/bjophthalmol-2011-300539. Epub 2011 Dec 1. PMID 22133988
- [Background] Chen DZ, Koh V, Sng C, Aquino MC, Chew P. Complications and outcomes of primary phacotrabeculectomy with mitomycin C in a multi-ethnic asian population. PLoS One. 2015 Mar 16;10(3):e0118852. doi: 10.1371/journal.pone.0118852. eCollection 2015. PMID 25775362
- [Background] Kung JS, Choi DY, Cheema AS, Singh K. Cataract surgery in the glaucoma patient. Middle East Afr J Ophthalmol. 2015 Jan-Mar;22(1):10-7. doi: 10.4103/0974-9233.148343. PMID 25624668
- [Background] Parikh HA, Bussel II, Schuman JS, Brown EN, Loewen NA. Coarsened Exact Matching of Phaco-Trabectome to Trabectome in Phakic Patients: Lack of Additional Pressure Reduction from Phacoemulsification. PLoS One. 2016 Feb 19;11(2):e0149384. doi: 10.1371/journal.pone.0149384. eCollection 2016. PMID 26895293
- [Background] Yang HS, Lee J, Choi S. Ocular biometric parameters associated with intraocular pressure reduction after cataract surgery in normal eyes. Am J Ophthalmol. 2013 Jul;156(1):89-94.e1. doi: 10.1016/j.ajo.2013.02.003. Epub 2013 Apr 28. PMID 23628350
- [Background] Lin SC, Masis M, Porco TC, Pasquale LR. Erratum: Predictors of Intraocular Pressure After Phacoemulsification in Primary Open-Angle Glaucoma Eyes with Wide Versus Narrower Angles (An American Ophthalmological Society Thesis). Trans Am Ophthalmol Soc. 2018 Jan 1;115:T6C1. eCollection 2017 Aug. PMID 29412193
- [Background] Baek SU, Kwon S, Park IW, Suh W. Effect of Phacoemulsification on Intraocular Pressure in Healthy Subjects and Glaucoma Patients. J Korean Med Sci. 2019 Jan 30;34(6):e47. doi: 10.3346/jkms.2019.34.e47. eCollection 2019 Feb 18. PMID 30787680
- [Background] O'Brien PD, Ho SL, Fitzpatrick P, Power W. Risk factors for a postoperative intraocular pressure spike after phacoemulsification. Can J Ophthalmol. 2007 Feb;42(1):51-5. PMID 17361241
- [Background] Potop V, Corbu C. The role of clear lens extraction in angle closure glaucoma. Rom J Ophthalmol. 2017 Oct-Dec;61(4):244-248. PMID 29516042
- [Background] Chen HY, Lin CL, Kao CH. Changes in glaucoma medication numbers after cataract and glaucoma surgery: A nationwide population-based study. Medicine (Baltimore). 2019 Jan;98(4):e14128. doi: 10.1097/MD.0000000000014128. PMID 30681574
- [Background] Vass C, Menapace R. Surgical strategies in patients with combined cataract and glaucoma. Curr Opin Ophthalmol. 2004 Feb;15(1):61-6. doi: 10.1097/00055735-200402000-00012. PMID 14743022
- [Background] Mercieca K, Shevade B, Anand N. Outcomes of combined phacoemulsification and deep sclerectomy: a 10-year UK single-centre study. Eye (Lond). 2015 Nov;29(11):1495-503. doi: 10.1038/eye.2015.163. Epub 2015 Sep 4. PMID 26337945
- [Background] Francis BA, Sarkisian SR, Tan JC (2017). Minimally invasive glaucoma surgery: A practical guide. 1st ed. New York: Thieme.
- [Background] Melamed S, Goldenfeld M, Cotlear D, Skaat A, Moroz I. High-intensity focused ultrasound treatment in refractory glaucoma patients: results at 1 year of prospective clinical study. Eur J Ophthalmol. 2015 Nov-Dec;25(6):483-9. doi: 10.5301/ejo.5000620. Epub 2015 May 13. PMID 25982212
- [Background] Mastropasqua R, Fasanella V, Mastropasqua A, Ciancaglini M, Agnifili L. High-Intensity Focused Ultrasound Circular Cyclocoagulation in Glaucoma: A Step Forward for Cyclodestruction? J Ophthalmol. 2017;2017:7136275. doi: 10.1155/2017/7136275. Epub 2017 Apr 22. PMID 28512580
- [Background] Giannaccare G, Vagge A, Sebastiani S, Urbini LE, Corazza P, Pellegrini M, Carmassi L, Bergamini F, Traverso CE, Campos EC. Ultrasound Cyclo-Plasty in Patients with Glaucoma: 1-Year Results from a Multicentre Prospective Study. Ophthalmic Res. 2019;61(3):137-142. doi: 10.1159/000487953. Epub 2018 May 16. PMID 29768281
- [Background] Gedde SJ, Schiffman JC, Feuer WJ, Herndon LW, Brandt JD, Budenz DL; Tube Versus Trabeculectomy Study Group. Three-year follow-up of the tube versus trabeculectomy study. Am J Ophthalmol. 2009 Nov;148(5):670-84. doi: 10.1016/j.ajo.2009.06.018. Epub 2009 Aug 11. PMID 19674729
- [Background] Francis BA, Berke SJ, Dustin L, Noecker R. Endoscopic cyclophotocoagulation combined with phacoemulsification versus phacoemulsification alone in medically controlled glaucoma. J Cataract Refract Surg. 2014 Aug;40(8):1313-21. doi: 10.1016/j.jcrs.2014.06.021. PMID 25088629
- [Background] Coleman DJ, Lizzi FL, Driller J, Rosado AL, Chang S, Iwamoto T, Rosenthal D. Therapeutic ultrasound in the treatment of glaucoma. I. Experimental model. Ophthalmology. 1985 Mar;92(3):339-46. doi: 10.1016/s0161-6420(85)34029-0. PMID 3991121
- [Background] De Gregorio A, Pedrotti E, Stevan G, Montali M, Morselli S. Safety and efficacy of multiple cyclocoagulation of ciliary bodies by high-intensity focused ultrasound in patients with glaucoma. Graefes Arch Clin Exp Ophthalmol. 2017 Dec;255(12):2429-2435. doi: 10.1007/s00417-017-3817-4. Epub 2017 Oct 17. PMID 29043438
- [Background] Pellegrini M, Sebastiani S, Giannaccare G, Campos EC. Intraocular inflammation after Ultrasound Cyclo Plasty for the treatment of glaucoma. Int J Ophthalmol. 2019 Feb 18;12(2):338-341. doi: 10.18240/ijo.2019.02.23. eCollection 2019. PMID 30809493
- [Background] Torky MA, Al Zafiri YA, Hagras SM, Khattab AM, Bassiouny RM, Mokbel TH. Safety and efficacy of ultrasound ciliary plasty as a primary intervention in glaucoma patients. Int J Ophthalmol. 2019 Apr 18;12(4):597-602. doi: 10.18240/ijo.2019.04.12. eCollection 2019. PMID 31024813
- [Background] Sun W, Yu CY, Tong JP. A review of combined phacoemulsification and endoscopic cyclophotocoagulation: efficacy and safety. Int J Ophthalmol. 2018 Aug 18;11(8):1396-1402. doi: 10.18240/ijo.2018.08.23. eCollection 2018. PMID 30140647
- [Background] Perez Bartolome F, Rodrigues IA, Goyal S, Bloch E, Lim WS, Alaghband P, Guajardo J, Jones S, Lim KS. Phacoemulsification plus endoscopic cyclophotocoagulation versus phacoemulsification alone in primary open-angle glaucoma. Eur J Ophthalmol. 2018 Mar;28(2):168-174. doi: 10.5301/ejo.5001034. PMID 29077182
- [Background] Hugo J, Matonti F, Beylerian M, Zanin E, Aptel F, Denis D. Safety and efficacy of high-intensity focused ultrasound in severe or refractory glaucoma. Eur J Ophthalmol. 2021 Jan;31(1):130-137. doi: 10.1177/1120672119874594. Epub 2019 Sep 25. PMID 31550914
- [Background] Heinz C, Zurek-Imhoff B, Koch J, Rosel M, Heiligenhaus A. Long-term reduction of laser flare values after trabeculectomy but not after cyclodestructive procedures in uveitis patients. Int Ophthalmol. 2011 Jun;31(3):205-10. doi: 10.1007/s10792-011-9440-1. Epub 2011 Mar 25. PMID 21437758
- [Background] Tan AM, Chockalingam M, Aquino MC, Lim ZI, See JL, Chew PT. Micropulse transscleral diode laser cyclophotocoagulation in the treatment of refractory glaucoma. Clin Exp Ophthalmol. 2010 Apr;38(3):266-72. doi: 10.1111/j.1442-9071.2010.02238.x. PMID 20447122
- [Background] Aquino MC, Barton K, Tan AM, Sng C, Li X, Loon SC, Chew PT. Micropulse versus continuous wave transscleral diode cyclophotocoagulation in refractory glaucoma: a randomized exploratory study. Clin Exp Ophthalmol. 2015 Jan-Feb;43(1):40-6. doi: 10.1111/ceo.12360. Epub 2014 Jun 21. PMID 24811050
- [Background] Liu GJ, Mizukawa A, Okisaka S. Mechanism of intraocular pressure decrease after contact transscleral continuous-wave Nd:YAG laser cyclophotocoagulation. Ophthalmic Res. 1994;26(2):65-79. doi: 10.1159/000267395. PMID 8196935
- [Background] Sousa DC, Ferreira NP, Marques-Neves C, Somers A, Vandewalle E, Stalmans I, Pinto LA. High-intensity Focused Ultrasound Cycloplasty: Analysis of Pupil Dynamics. J Curr Glaucoma Pract. 2018 Sep-Dec;12(3):102-106. doi: 10.5005/jp-journals-10028-1253. PMID 31354201
- [Background] Rivero-Santana A, Perez-Silguero D, Perez-Silguero MA, Encinas-Pisa P. Pupil Ovalization and Accommodation Loss after High-intensity Focused Ultrasound Treatment for Glaucoma: A Case Report. J Curr Glaucoma Pract. 2019 May-Aug;13(2):77-78. doi: 10.5005/jp-journals-10078-1256. PMID 31564798
- [Background] Bolek B, Wylegala A, Wylegala E. Ultrasound ciliary plasty in glaucoma treatment: A long-term follow-up study. Acta Ophthalmol. 2023 May;101(3):293-300. doi: 10.1111/aos.15290. Epub 2022 Nov 30. PMID 36448501
- [Background] Deb-Joardar N, Reddy KP. Application of high intensity focused ultrasound for treatment of open-angle glaucoma in Indian patients. Indian J Ophthalmol. 2018 Apr;66(4):517-523. doi: 10.4103/ijo.IJO_1024_17. PMID 29582811
- [Derived] Torky MA, Alzafiri YA, Abdelhameed AG, Awad EA. Phaco-UCP; combined phacoemulsification and ultrasound ciliary plasty versus phacoemulsification alone for management of coexisting cataract and open angle glaucoma: a randomized clinical trial. BMC Ophthalmol. 2021 Jan 21;21(1):53. doi: 10.1186/s12886-021-01818-5. PMID 33478426